CLINICAL TRIAL: NCT04228887
Title: Effects of Inspiratory Muscle Training on Postural Stability, Mobility, Activities of Daily Living, Quality of Life and Respiratory Function in Patients With Parkinson's Disease
Brief Title: Effects of Inspiratory Muscle Training in Patients With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BezmialemVU27
Record Dates: First submitted 2019-08-05; First posted 2020-01-14 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; Inspiratory Muscle Training; Balance Training
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): The control group will be receive 45 minutes training sessions 3 times a week for 8 weeks; 2 days a week for home based balance training and 1 day for supervisory training with Bio-Dex Balance-System ®.
  Interventions: Diagnostic Test: Respiratory Muscle Strength; Device: Balance Training
- Training Group (Active Comparator): The training group will receive inspiratory muscle training; 15 minutes sessions 5 times a week for 8 weeks in addion to balance training same as control.
  Interventions: Diagnostic Test: Respiratory Muscle Strength; Device: Balance Training; Device: Inspiratory Muscle Training

INTERVENTIONS:
Diagnostic Test: Respiratory Muscle Strength — Respiratory muscle strengths will evalueted with inspiratory and expiratory mouth pressure devices.
Device: Balance Training — Balance training will provide with Biodex® Balance Training System
Device: Inspiratory Muscle Training — 15 minutes twice a day, 5 times a week for 8 week with Threshold IMT device
  Arms: Training Group

SUMMARY:
In this study investigators will examine the effects of inspiratory muscle training and balance training in patients with Parkinson's Disease

DETAILED DESCRIPTION:
Parkinson's Disease (PD) is the most common type of Parkinsonism and mainly due to degeneration of basal ganglions and substantia nigra occurs. Balance disorders are one of the common problems in patients with Parkinson's disease. These balance disorders; loss of postural reflexes, insufficiency in postural adjustments, rigidity in the trunk and extremities, and many disorders such as akinesia. Because of balance disorders in patients with PD, increase in addiction to daily life activities, causes physical disability. In the case of PD pulmonary problems may be the leading cause of mortality and mortality. Respiratory symptoms in these patients cause problems in weakness, swallowing, coughing, voice and speech functions. When the investigators look at the current literature, the effect of balance and respiration on Parkinson's patients is found to be seperately but their effect on each other is not sufficiently emphasized. For this reason, the researchers' aim to investigate balance and postural control in patients with Parkinson's disease and to increase the strength of respiratory muscles and to improve balance and postural control.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Parkinson'S Disease
* Ages between 60 and 85 years
* Grades 1 to 3 according to Modified Hoehn-Yahr Scale

Exclusion Criteria:

* Lung surgery or diagnosed lung disease history
* Dementia
* Having a orthopedic disorder which may affect balance and/or mobility
* Severe dyskinesia and cognition problems

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-05-04 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Inspiratory Muscle Strength | Change from baselines to final evaluation at 8th weeks
  Maximal inspiratory pressure (MIP) is the most widely used measure of respiratory muscle strength in patients with suspected respiratory muscle weakness. It is determined by measuring upper airway pressure (mouth for outpatients and trachea for intubated or tracheostomized patients) during a maximal voluntary inspiratory effort. The measured pressure is a composite of the pressure generated by the inspiratory muscles and the elastic recoil pressure of the lungs and chest wall.
Respiratory Function- Forced Vital Capasity (FVC) | Change from baselines to final evaluation at 8th weeks
  Forced vital capacity (FVC) is the total amount of air exhaled during the FEV test. FVC can also help doctors assess the progression of lung disease and evaluate the effectiveness of treatment.
Respiratory Function- Forced Expiratory Volume in 1 second | Change from baselines to final evaluation at 8th weeks
  Forced expiratory volume (FEV) measures how much air a person can exhale during a forced breath. Forced expiratory volume and forced vital capacity are lung function tests that are measured during spirometry. Forced expiratory volume is the most important measurement of lung function. It is used to:
  Diagnose obstructive lung diseases such as asthma and chronic obstructive pulmonary disease (COPD). A person who has asthma or COPD has a lower FEV1 result than a healthy person.
  See how well medicines used to improve breathing are working. Check if lung disease is getting worse. Decreases in the FEV1 value may mean the lung disease is getting worse.
Respiratory Function- Peak Expiratory Flow | Change from baselines to final evaluation at 8th weeks
  The peak expiratory flow (PEF), also called peak expiratory flow rate (PEFR), is a person's maximum speed of expiration, as measured with a peak flow meter, a small, hand-held device used to monitor a person's ability to breathe out air.
Postural Control and Balance | Change from baselines to final evaluation at 8th weeks
  Biodex Balance System evaluations
Parkinson's Status- Unified Parkinson's Disease Rating Scale | Change from baselines to final evaluation at 8th weeks
  The UPDRS scale refers to Unified Parkinson Disease Rating Scale, and it is a rating tool used to gauge the course of Parkinson's disease in patients. The UPDRS scale includes series of ratings for typical Parkinson's symptoms that cover all of the movement hindrances of Parkinson's disease. The UPDRS scale consists of the following five segments: 1) Mentation, Behavior, and Mood, 2) ADL, 3) Motor sections, 4) Modified Hoehn and Yahr Scale, and 5) Schwab and England ADL scale. Each answer to the scale is evaluated by a medical professional that specializes in Parkinson's disease during patient interviews.

SECONDARY OUTCOMES:
Mobility Status- Rivermead mobility index | Change from baselines to final evaluation at 8th weeks
  The Rivermead Mobility Index assesses functional mobility in gait, balance and transfers. The Rivermead Mobility Index is appropriate for a range of disabilities that include anything from being bedridden to being able to run 15 items:
  14-self-reported items
  1 direct observation item Items progress in difficulty Items are coded as either 0 or 1, depending on whether the patient can complete the task according to specific instructions Items receive a score of 0 for a "No" response and 1 for a "Yes" response Total scores are determined by summing the points for all items A maximum of 15 points is possible; higher scores indicate better mobility performance A score of "0" indicates an inability to perform any of the activities on the measure
Quality of Life Parameter-Nottingham Health Profile | Change from baselines to final evaluation at 8th weeks
  The Nottingham Health Profile is intended for primary health care, to provide a brief indication of a patient's perceived emotional, social and physical health problems. Breakdown of questionaire
  (1) Part I: 38 questions in 6 subareas, with each question assigned a weighted value; the sum of all weighted values in a given subarea adds up to 100
  * energy level (EL): 3
  * pain (P): 8
  * emotional reaction (ER): 9
  * sleep (S): 5
  * social isolation (SI): 5
  * physical abilities (PA): 8
Activities of Daily Living-Barthel | Change from baselines to final evaluation at 8th weeks
  The Barthel Scale/Index (BI) is an ordinal scale used to measure performance in activities of daily living (ADL). Ten variables describing ADL and mobility are scored, a higher number being a reflection of greater ability to function independently following hospital discharge.Time taken and physical assistance required to perform each item are used in determining the assigned value of each item. The Barthel Index measures the degree of assistance required by an individual on 10 items of mobility and self care ADL.

CONTACTS AND LOCATIONS:
Overall Officials: Hülya N Gürses, Prof, Study Director — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No